CLINICAL TRIAL: NCT02132936
Title: LEO 90100 Aerosol Foam Compared to Calcipotriol Plus Betamethasone Dipropionate Gel in Subjects With Psoriasis Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LP0053-1003
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2016-07

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Gels

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LEO 90100 (Experimental): LEO 90100 aerosol foam, containing calcipotriol (as hydrate) 50 mcg/g and betamethasone 0.5 mg/g (as dipropionate), 60 g per can, applied once daily up to 12 weeks
  Interventions: Drug: LEO 90100 aerosol foam
- Aerosol foam vehicle (Placebo Comparator): Aerosol foam vehicle, 60 g per can, applied once daily for up to 12 weeks
  Interventions: Drug: Aerosol foam vehicle
- Calcipotriol BDP gel (Active Comparator): Calcipotriol BDP gel, containing calcipotriol (as hydrate) 50 mcg/g and betamethasone 0.5 mg/g (as dipropionate), 60 g per bottle, applied once daily up to 12 weeks
  Interventions: Drug: Calcipotriol BDP gel
- Gel vehicle (Placebo Comparator): Gel vehicle, 60 g per bottle, applied once daily up to 12 weeks
  Interventions: Drug: Gel vehicle

INTERVENTIONS:
Drug: LEO 90100 aerosol foam
  Arms: LEO 90100
Drug: Aerosol foam vehicle
  Arms: Aerosol foam vehicle
Drug: Calcipotriol BDP gel
  Arms: Calcipotriol BDP gel
Drug: Gel vehicle
  Arms: Gel vehicle

SUMMARY:
The purpose is to compare the efficacy of treatment with LEO 90100 at Week 4 to that of calcipotriol plus betamethasone dipropionate (BDP) gel at Week 8 in subjects with psoriasis vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Psoriasis vulgaris on the trunk and/or limbs (excluding psoriasis on the genitals and skin folds) involving 2-30% of the Body Surface Area (BSA)
* A Physician's Global Assessment of disease severity (PGA) of at least mild on trunk and limbs
* A modified Psoriasis Area Severity Index (PASI) score of at least 2 on the trunk and limbs.

Exclusion Criteria:

* Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis
* Systemic treatment with biological therapies, whether marketed or not, with a possible effect on psoriasis vulgaris within the following time periods prior to randomisation:

  * etanercept - within 4 weeks prior to randomisation
  * adalimumab, infliximab - within 8 weeks prior to randomisation
  * ustekinumab - within 16 weeks prior to randomisation
  * other products - within 4 weeks/5 half-lives prior to randomisation (whichever is longer)
* Systemic treatment with all other therapies with a possible effect on psoriasis vulgaris (e.g. corticosteroids, retinoids, methotrexate, ciclosporin and other immunosuppressants within 4 weeks prior to randomisation)
* Subjects who have received treatment with any non-marketed drug substance (i.e. a drug which has not yet been made available for clinical use following registration) within 4 weeks/5 half-lives (whichever is longer) prior to randomisation.
* Psoralen combined with Ultraviolet A (PUVA) therapy within 4 weeks prior to randomisation
* Ultraviolet B (UVB) therapy within 2 weeks prior to randomisation
* Topical anti-psoriatic treatment on the trunk and limbs (except for emollients) within 2 weeks prior to randomisation
* Topical treatment on the face, scalp and skin folds with corticosteroids, vitamin D analogues or prescription shampoos within 2 weeks prior to randomisation
* Females who are pregnant, wishing to become pregnant during the trial or are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Dermatologie, Hôspital Larrey, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paul C, Stein Gold L, Cambazard F, Kalb RE, Lowson D, Bang B, Griffiths CE. Calcipotriol plus betamethasone dipropionate aerosol foam provides superior efficacy vs. gel in patients with psoriasis vulgaris: randomized, controlled PSO-ABLE study. J Eur Acad Dermatol Venereol. 2017 Jan;31(1):119-126. doi: 10.1111/jdv.13859. Epub 2016 Aug 17. PMID 27531752
- [Derived] Veverka KA, Hansen JB, Yaloumis M, Kircik L, Stein Gold L. Calcipotriene Plus Betamethasone Dipropionate Foam for Mild Psoriasis: Pooled Results from Three Randomized Trials. J Drugs Dermatol. 2021 Aug 1;20(8):822-828. doi: 10.36849/JDD.5743. PMID 34397196
- [Derived] Iversen L, Kurvits M, Snel-Prento AM, Menter A. Calcipotriol/Betamethasone Dipropionate Cutaneous Foam Treatment for Psoriasis in Patients With BSA 5-15% and PGA >/= 3: Post-Hoc Analysis From Three Randomized Controlled Trials. Dermatol Ther (Heidelb). 2020 Oct;10(5):1111-1120. doi: 10.1007/s13555-020-00419-2. Epub 2020 Aug 12. PMID 32785881
- [Derived] Paul C, Leonardi C, Menter A, Reich K, Gold LS, Warren RB, Moller A, Lebwohl M. Calcipotriol Plus Betamethasone Dipropionate Aerosol Foam in Patients with Moderate-to-Severe Psoriasis: Sub-Group Analysis of the PSO-ABLE Study. Am J Clin Dermatol. 2017 Jun;18(3):405-411. doi: 10.1007/s40257-017-0258-0. PMID 28236223
- Available data/document: Clinical Study Report — https://www.leopharmatrials.com/en — Clinical Trials at LEO Pharma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 30-Jun-2014 Last Subject Last Visit: 04-Mar-2015
Pre-assignment Details: A total of 504 subjects were enrolled, 41 enrolled subjects were not randomised. 463 subjects were randomised as follows: 185 subjects to LEO 90100, 188 to calcipotriol BDP gel, 47 to foam vehicle, and 43 to gel vehicle
Period: Overall Study
Arm/Group | LEO 90100 | Aerosol Foam Vehicle | Calcipotriol BDP Gel | Gel Vehicle
Started | 185 | 47 | 188 | 43
Completed | 175 | 38 | 174 | 29
Not Completed | 10 | 9 | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- LEO 90100: LEO 90100 aerosol foam, containing calcipotriol (as hydrate) 50 mcg/g and betamethasone 0.5 mg/g (as dipropionate), 60 g per can, applied once daily up to 12 weeks
  LEO 90100 aerosol foam
- Aerosol Foam Vehicle: Aerosol foam vehicle, 60 g per can, applied once daily for up to 12 weeks
  Aerosol foam vehicle
- Calcipotriol BDP Gel: Calcipotriol BDP gel, containing calcipotriol (as hydrate) 50 mcg/g and betamethasone 0.5 mg/g (as dipropionate), 60 g per bottle, applied once daily up to 12 weeks
  Calcipotriol BDP gel
- Gel Vehicle: Gel vehicle, 60 g per bottle, applied once daily up to 12 weeks
  Gel vehicle
- Total: Total of all reporting groups
Arm/Group | LEO 90100 | Aerosol Foam Vehicle | Calcipotriol BDP Gel | Gel Vehicle | Total
Number analyzed (Participants) | 185 | 47 | 188 | 43 | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (14.5) | 54.6 (14.2) | 54.5 (14.9) | 51.9 (15.5) | 54.1 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 18 | 74 | 17 | 168
  Male | 126 | 29 | 114 | 26 | 295

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success According to the PGA
Description: To compare the efficacy of treatment of LEO 90100 at Week 4 to that of calcipotriol BDP gel at Week 8 in subjects with psoriasis vulgaris.
  Five-point assessment (clear, almost clear, mild, moderate, and severe) was made for the severity of psoriasis vulgaris on the trunk and limbs at all on-treatment visits using Physician's Global Assessment of Disease Severity (PGA).
  'Treatment success' was defined as achieving 'clear' or 'almost clear' for subjects with at least 'moderate' disease at baseline and 'clear' for subjects with 'mild' disease at baseline.
Time Frame: 4 Weeks for LEO 90100 and 8 weeks for calcipotriol BDP gel
Measure: Number; unit: percentage of subjects
Arm/Group | LEO 90100 | Calcipotriol BDP Gel
Number analyzed (Participants) | 185 | 188
percentage of subjects | 38.3 | 22.5
Statistical Analysis 1: Comparison: LEO 90100 vs Calcipotriol BDP Gel; Mantel-Haenszel odds of treatment success in LEO 90100 group relative to calcipotriol BDP gel group, adjusted for pooled centre and baseline PGA. Multiple imputation was used to handle missing PGA values; Test type: Superiority or Other; p < 0.001, Mantel Haenszel; Odds Ratio (OR) = 2.55, 95% CI 2-sided [1.46 to 4.46]

2. Secondary Outcome: Subjects With PASI 75 at Week 4 for LEO 90100 and at Week 8 for Calcipotriol BDP Gel.
Description: Subjects with PASI 75 (a 75% reduction in the modified Psoriasis Area and Severity Index) at Week 4 for LEO 90100 and at Week 8 for calcipotriol BDP gel.
Time Frame: Week 4 for LEO 90100; Week 8 for calcipotriol BDP gel
Measure: Number; unit: percentage of subjects
Arm/Group | LEO 90100 | Calcipotriol BDP Gel
Number analyzed (Participants) | 185 | 188
percentage of subjects | 52.1 | 34.6
Statistical Analysis 1: Comparison: LEO 90100 vs Calcipotriol BDP Gel; Mantel-Haenszel odds of having PASI 75 in LEO 90100 group relative to calcipotriol BDP gel group, adjusted for pooled centre and baseline PGA. Multiple imputation was used to handle missing data; Test type: Superiority or Other; p = 0.001, Mantel Haenszel; Odds Ratio (OR) = 2.18, 95% CI 2-sided [1.37 to 3.47]

3. Secondary Outcome: Time to 'Treatment Success' According to PGA.
Description: Time to treatment success was calculated as the number of weeks from baseline to the visit where the subject first achieved treatment success.
  'Treatment success' was defined as achieving 'clear' or 'almost clear' for subjects with at least 'moderate' disease at baseline and 'clear' for subjects with 'mild' disease at baseline.
Time Frame: From Baseline to Week 12
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | LEO 90100 | Calcipotriol BDP Gel
Number analyzed (Participants) | 185 | 188
weeks | 6 [4 to NA] — Upper quartile could not be estimated as less than 75% of subjects achieved treatment success. | NA [6 to NA] — Median could not be estimated for the calcipotriol BDP gel group as less than 50% of subjects achieved treatment success. Upper quartile could not be estimated as less than 75% of subjects achieved treatment success.
Statistical Analysis 1: Comparison: LEO 90100 vs Calcipotriol BDP Gel; Test type: Superiority or Other; p < 0.001, Log Rank

4. Secondary Outcome: Change in Itch as Assessed on a VAS Scale (LEO 90100 vs. the Foam Vehicle Group).
Description: Maximum itch during the previous 24 hours was assessed on a Visual Analogue Scale (VAS) - range from 0 (no itch at all) to 100 mm (worst itch one could imagine).
Time Frame: Baseline to Week 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LEO 90100 | Aerosol Foam Vehicle
Number analyzed (Participants) | 185 | 47
units on a scale | -30.5 [-33.4 to -27.5] | -15.9 [-21.3 to -10.5]
Statistical Analysis 1: Comparison: LEO 90100 vs Aerosol Foam Vehicle; Mean change in itch adjusted for pooled centre, baseline PGA and baseline itch. Multiple imputation used for missing data; Test type: Superiority or Other; p < 0.001, ANCOVA

5. Secondary Outcome: Change in Itch as Assessed on a VAS Scale From Baseline to Week 4 (LEO 90100) vs. Week 8 (Calcipotriol BDP Gel).
Description: Maximum itch during the previous 24 hours was assessed on a Visual Analogue Scale - range from 0 (no itch at all) to 100 mm (worst itch one could imagine).
Time Frame: Baseline to Week 4; Baseline to Week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | LEO 90100 | Calcipotriol BDP Gel
Number analyzed (Participants) | 185 | 188
units on a scale | -30.5 [-33.4 to -27.5] | -28.5 [-31.4 to -25.6]
Statistical Analysis 1: Comparison: LEO 90100 vs Calcipotriol BDP Gel; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.33, ANCOVA

ADVERSE EVENTS:
Time Frame: Day 0 until week 12
Arm/Group | LEO 90100 | Aerosol Foam Vehicle | Calcipotriol BDP Gel | Gel Vehicle
Serious Adverse Events (participants affected / at risk) | 4/185 | 0/47 | 3/188 | 1/43
Other Adverse Events (participants affected / at risk) | 62/185 | 25/47 | 60/188 | 28/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 90100 (N=185) | Aerosol Foam Vehicle (N=47) | Calcipotriol BDP Gel (N=188) | Gel Vehicle (N=43)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 (N=185) | Aerosol Foam Vehicle (N=47) | Calcipotriol BDP Gel (N=188) | Gel Vehicle (N=43)
Nasopharyngitis (Infections and infestations) | 7 (7) | 0 (0) | 4 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 1 (1) | 9 (9) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 6 (6) | 0 (0) | 5 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 3 (3) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1) | 2 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 7 (8) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 7 (7) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Intertrigo candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Application site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.